CLINICAL TRIAL: NCT00216632
Title: Treatment Success in Patients Requiring Treatment Change From Olanzapine to Risperidone Long Acting Injectable (TRESOR)
Brief Title: A Study of Treatment Success in Changing From Olanzapine to Long-acting Injectable Risperidone (RISPERDAL® CONSTA™)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003211
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Schizophrenia, Schizoaffective disorder; antipsychotic agents; long-acting risperidone; intramuscular injection
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to evaluate the maintained effectiveness of long-acting injectable risperidone (RISPERDAL® CONSTA™) compared with the previous treatment with oral olanzapine in non-acute subjects with schizophrenia or schizoaffective disorder considered in need of a therapy change.

DETAILED DESCRIPTION:
Although many schizophrenia patients currently take oral antipsychotic medications, it is estimated that up to 75% of them have difficulty adhering to the daily oral regimen. Long-acting injectable formulations may eliminate the need for daily medication and enhance patient compliance with the treatment regimen. In addition, transitioning to a different antipsychotic drug is at times a necessary step in the clinical management of patients with schizophrenia due to different reasons, including insufficient response and poor tolerability. This is an open-label, non-randomized study of a formulation of risperidone (RISPERDAL® CONSTA™) (coated microspheres) injected into the muscle at week intervals over 6 months in patients with schizophrenia or schizoaffective disorder. During the first 3 weeks, oral olanzapine treatment is continued to provide therapy until the risperidone long-acting injectable reaches effective drug levels. The oral olanzapine treatment is tapered off within 1 week for one group of patients and within 3 weeks for another group. Assessments of effectiveness include the Positive and Negative Syndrome Scale (PANSS), overall severity of illness measured by the Clinical Global Impression (CGI) scale, and quality of life evaluated by the SF-36 questionnaire. Safety evaluations include incidence of adverse events through out the study and Extrapyramidal Symptom Rating Scale (ESRS), clinical laboratory tests (biochemistry, hematology, and urinalysis), and physical exams, including body weight, at specified intervals. The study hypothesis is that changing to treatment every 2 weeks with long-acting risperidone will provide a maintained effectiveness patients with schizophrenia or schizoaffective disorder and will be generally well-tolerated Risperidone, long-acting formulation for intramuscular injection (25 milligrams[mg]) every 2 weeks for 6 months. Investigator may adjust dosage to 37.5mg or 50mg (maximum) or supplement risperidone injections with risperidone tablets (2mg maximum), according to symptoms and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder according to criteria of Diagnostic and StatisticalManual of Mental Diseases, 4th edition (DSM-IV)
* patients must have been symptomatically non-acute on a stable dose of olanzapine the last month before the screening visit
* patients must be currently treated with oral olanzapine at doses stable for the last month and willing to switch to long-acting injectable risperidone for one of the following reasons: insufficient treatment response, adverse events, compliance issues, or patient's request.

Exclusion Criteria:

* Patients not treated with effective doses of olanzapine (acc. to SmPC) prior to study initiation
* known hypersensitivity, intolerance, or unresponsiveness to risperidone
* history of drug allergy or neuroleptic malignant syndrome, a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness
* tardive dyskinesia, a complication of neuroleptic therapy involving involuntary movements of facial muscles
* pregnant or nursing females, or those lacking adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2005-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total Positive and Negative Syndrome Scale (PANSS) score at the end of the treatment period (6 months).

SECONDARY OUTCOMES:
Changes from baseline to end of treatment in Clinical Global Impression-Severity of Illness, Quality of Life SF-36, patient satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Derived] Rosa F, Schreiner A, Thomas P, Sherif T. Switching patients with stable schizophrenia or schizoaffective disorder from olanzapine to risperidone long-acting injectable. Clin Drug Investig. 2012 Apr 1;32(4):267-79. doi: 10.2165/11599080-000000000-00000. PMID 22339430